CLINICAL TRIAL: NCT02688270
Title: A Double-blinded Crossover Study of Topical Formulation of Nitroglycerine, Vascana®, Versus Matching Vehicle in the Subjective and Physiologic Responses to Controlled Cold Challenge in Subjects With Raynaud's Phenomenon (RP) Secondary to Connective Tissue Disease
Brief Title: Efficacy and Safety of Vascana® in Subjects With Secondary Raynaud's Phenomenon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Covis Pharma S.à.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VAS-014-001
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Results first posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Raynaud's Phenomenon Secondary to Connective Tissue Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Sequence A (Experimental): Vascana® (0.9% nitroglycerin cream), Vehicle cream, Vascana® (0.9% nitroglycerin cream), Vehicle cream
  Interventions: Drug: Vascana (0.9% nitroglycerin cream); Drug: Vehicle Cream (placebo)
- Treatment Sequence B (Experimental): Vascana® (0.9% nitroglycerin cream), Vehicle cream, Vehicle cream, Vascana® (0.9% nitroglycerin cream)
  Interventions: Drug: Vascana (0.9% nitroglycerin cream); Drug: Vehicle Cream (placebo)
- Treatment Sequence C (Experimental): Vehicle cream, Vascana® (0.9% nitroglycerin cream), Vehicle cream, Vascana® (0.9% nitroglycerin cream)
  Interventions: Drug: Vascana (0.9% nitroglycerin cream); Drug: Vehicle Cream (placebo)
- Treatment Sequence D (Experimental): Vehicle cream, Vascana® (0.9% nitroglycerin cream), Vascana® (0.9% nitroglycerin cream), Vehicle cream
  Interventions: Drug: Vascana (0.9% nitroglycerin cream); Drug: Vehicle Cream (placebo)

INTERVENTIONS:
Drug: Vascana (0.9% nitroglycerin cream) — Study drug administered topically
Drug: Vehicle Cream (placebo) — Vehicle administered topically

SUMMARY:
The purpose of this study is to determine the ability of Vascana (0.9% nitroglycerin topical cream) to treat and prevent the symptoms experienced by subject's with Raynaud's Phenomenon. The symptoms of this disease include pain, tingling, and numbness in the fingers of the affected hand or hands.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written consent prior to any study-specific evaluation
2. Males and females aged 18 years to 75 years, inclusive
3. A clinical diagnosis of secondary Raynaud's Phenomenon (defined as Raynaud's Phenomenon (RP) significant enough to cause a patient to modify daily behavior) as determined by a history of cold sensitivity with pain, numbness, and/or tingling along with pallor or cyanosis of the fingers, or by such an event observed by the study physician and a diagnosis of a disease state known to be associated with RP. Secondary RP may be due to scleroderma, systemic lupus erythematosus, mixed connective tissue disease, or other connective tissue diseases
4. Agree to apply the study drug to their fingers as specified in the protocol
5. Agree to the controlled cold exposures as described in the protocol
6. Willing to discontinue current vasodilator therapies used specifically for the treatment of Raynaud's
7. Agree not to use any other investigational medications or approved or unapproved therapies to treat RP and its symptoms while participating in this study. Such medications include, but are not limited to: other dosages forms of nitroglycerin, eg, isosorbide dinitrate, fenoldopam mesylate, milrinone lactate, nifedipine, diltiazem, felodipine, nimodipine, nisoldipine, fluoxetine, pregabalin, and verapamil. Use of phosphodiesterase 5 inhibitors (eg, sildenafil, tadalafil, vardenafil) is excluded unless being used intermittently for male erectile dysfunction and not taken within 48 hours of scheduled study drug dosing
8. Negative urine pregnancy test for women of child-bearing potential prior to the first study treatment and who agree to use effective contraception throughout the study
9. Able to comply with all study requirements

Exclusion Criteria:

1. Past history of RP attacks of sufficient severity as to require inpatient hospitalization
2. Presence of an active digital ulcer defined as a painful ulcer with visible depth and loss of epithelialization. Ulcers covered with eschar wherein depth and epithelialization cannot be judged are said to be "indeterminant" and are not exclusionary.
3. Raynaud's Phenomenon secondary to non-connective tissue disorders including thromboangiitis obliterans (Buerger's disease), hemorheologic disorders, major arterial occlusive disease, past exposure to vasopathic agents (including vinblastine, cis platinum, and bleomycin), ongoing therapy with vasoconstrictive agents (eg, beta-blockers), and past frostbite injury amongst others. Subjects with hepatitis C should also be excluded.
4. Patients diagnosed with pulmonary arterial hypertension requiring specific therapy.
5. Concurrently using any nitrate medication or medications known to interact with nitroglycerin such as sildenafil, and other treatments for erectile dysfunction beyond screening. Subjects may participate in the study once these drugs have been discontinued for at least 5 half-lives
6. Concurrently using any medication or device which might interfere with the study medication (including RP therapies, drugs used for hypertension, arrhythmia, depression, and pain), specifically calcium channel blockers and the compounds listed in prohibited concomitant medications beyond screening, unless such medication is required for a condition other than Raynaud's. Subjects may participate in the study once these drugs have been discontinued for at least 5 half-lives.
7. Known allergy to nitroglycerin or common topical cream ingredients
8. History of migraine, cluster, or vascular headaches, or chronic pain (defined as pain of 3-hour duration or longer on a daily basis) with greater intensity than the pain associated with RP or other chronic pain condition in their fingers
9. Any unstable medical problem or any current medical condition that, in the judgment of the investigator, would contraindicate the administration of the study medication, interfere with the study evaluations, or interfere with the subject's ability to comply with the study protocol
10. Cognitive or language difficulties that would impair completion of the symptom assessment instruments
11. Within the past 3 months, have had a myocardial infarction, uncontrolled congestive heart failure, unstable angina, uncontrolled hypotension, or uncontrolled hypertension (defined as subjects not being treated medically to control these conditions)
12. Participated in a study of any investigational drug within 4 weeks prior to visit 1
13. Screening laboratory values are 20% or more from the upper or lower limit of normal and that are considered to be clinically significant to the investigator
14. Had major abdominal, thoracic, or vascular surgery within 6 months of visit 1
15. Pregnant or nursing women
16. Women of childbearing potential who are unable or unwilling to comply with the contraceptive requirements during the study period
17. History of relevant drug and/or food allergies that resulted in a systemic reaction that required medical treatment
18. History of alcohol abuse or drug addiction which in the estimation of the principal investigator would affect the subjects ability to participate in the study
19. Consumption of alcohol on day before a visit and day of the visit.
20. Consumption of two or more alcoholic beverages on a daily basis.
21. Use of tobacco products of any type and at any level in the preceding 6 months and for the duration of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple investigational sites, Multiple Locations, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Sequence A | Treatment Sequence B | Treatment Sequence C | Treatment Sequence D
Started | 16 | 16 | 17 | 16
Completed | 16 | 16 | 17 | 16
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence A | Treatment Sequence B | Treatment Sequence C | Treatment Sequence D | Total
Number analyzed (Participants) | 16 | 16 | 17 | 16 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (13.37) | 53.8 (11.42) | 52.1 (16.24) | 47.7 (13.34) | 51.4 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 16 | 15 | 60
  Male | 2 | 1 | 1 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 17 | 16 | 65

OUTCOME MEASURES:

1. Primary Outcome: Raynaud's Symptom Severity (Change From Baseline)
Description: Change from baseline to visit 6 in peak Main Raynaud's Symptom (MRS) severity. Raynaud's symptoms will be assessed separately using a 0 to100-mm Visual Analog Scale (VAS) for pain, numbness, and tingling where 0 mm = no symptom and 100 mm = most severe symptom.
Time Frame: 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Vascana: Vascana (0.9% nitroglycerin cream): Study drug administered topically
- Vehicle Cream: Vehicle Cream (placebo): Vehicle administered topically
Arm/Group | Vascana | Vehicle Cream
Number analyzed (Participants) | 65 | 65
score on a scale | -20.19 [-26.63 to -13.75] | -18.63 [-25.07 to -12.19]

2. Primary Outcome: Raynaud's Symptom Severity (Percentage of Responders)
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Vascana | Vehicle Cream
Number analyzed (Participants) | 65 | 65
Participants | 37 | 29

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Vascana | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 17/65 | 16/65
Other Adverse Events (participants affected / at risk) | 1/17 | 3/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vascana (N=65) | Vehicle Cream (N=65)
Blood Pressure Increased (Vascular disorders) | 8 (8) | 7 (7)
Nervous System Disorders (Nervous system disorders) | 1 (1) | 4 (4)
General disorders and administration site conditions (General disorders) | 3 (3) | 1 (1)
Infections and infestations (Infections and infestations) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 3 (3)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vascana (N=17) | Vehicle Cream (N=16)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Blood Pressure Increased (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No